CLINICAL TRIAL: NCT03508739
Title: Glucagon-like Peptide-1 Metabolism in the Setting of Acute Neprilysin Inhibition
Brief Title: Glucagon-like Peptide-1 Metabolism and Acute Neprilysin Inhibition
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: We do not have active funding at this time.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jessica R.Wilson, MD, MS, Instructor in Medicine Division of Endocrinology, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 828731
Record Dates: First submitted 2017-11-07; First posted 2018-04-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetic; Hypertension; Elevated Blood Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Hypertension | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: prospective randomized, double-blind, crossover study, mechanistic/ translational study (not to change labeling or marketing, not classic phase 3 or 4 study), IND exempt
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM 1: randomization order AB (Experimental): Subjects will present for a baseline mixed meal study day 1 (no medication). Next they will be randomized to sacubitril/valsartan 200mg po and then valsartan 160 mg po with each medication given on study day 2 and 3, respectively (order AB). At each study day, subjects will present after fasting and receive blinded study medication on study days 2 and 3. After an IV is placed, neprilysin activity will be measured at baseline. Two hours later, subjects will have neprilysin activity collected again as well as baseline insulin, glucose, GLP-1, and triglycerides. Following this, subjects will ingest a mixed meal. Blood samples for insulin, glucose, GLP-1, and triglycerides will be collected after the meal for four hours total. Blood pressure and heart rate will be monitored.
  Interventions: Drug: Sacubitril/Valsartan 200mg (blinded); Drug: Valsartan 160mg (blinded)
- ARM 2: randomization order BA (Experimental): Subjects will present for a baseline mixed meal study day 1 (no medication). Next they will be randomized to sacubitril/valsartan 200mg po and then valsartan 160 mg po with each medication given on study day 2 and 3, respectively (order BA). At each study day, subjects will present after fasting and receive blinded study medication on study days 2 and 3. After an IV is placed, neprilysin activity will be measured at baseline. Two hours later, subjects will have neprilysin activity collected again as well as baseline insulin, glucose, GLP-1, and triglycerides. Following this, subjects will ingest a mixed meal. Blood samples for insulin, glucose, GLP-1, and triglycerides will be collected after the meal for four hours total. Blood pressure and heart rate will be monitored.
  Interventions: Drug: Sacubitril/Valsartan 200mg (blinded); Drug: Valsartan 160mg (blinded)

INTERVENTIONS:
Drug: Sacubitril/Valsartan 200mg (blinded) — study day 2 for AB and study day 3 for BA
  Other Names: Entresto
Drug: Valsartan 160mg (blinded) — study day 3 for AB and study day 2 for BA
  Other Names: Diovan

SUMMARY:
Type 2 diabetes is common, increases in prevalence with age, and patients with diabetes have an increased risk of cardiovascular disease. A relatively new cardiovascular medication currently used for the treatment of heart failure in the United States inhibits an enzyme that breaks down a variety of signaling hormones. This clinical trial tests if it may also be a target for the treatment of diabetes by decreasing the breakdown of a hormone that increases insulin release after a meal.

DETAILED DESCRIPTION:
This study will test the hypothesis that neprilysin inhibition with sacubitril/valsartan will increase endogenous glucagon-like peptide-1 (GLP-1) after a mixed meal compared to valsartan. The primary statistical analysis will be within subject comparison (paired t-test or nonparametric equivalent) of area under the curve intact GLP-1 after the meal during sacubitril/valsartan compared to valsartan. Neprilysin inhibition may be a new drug target for the treatment of type 2 diabetes by increasing intact GLP-1 and may be of particular benefit to individuals with increased risk of hypoglycemia and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-80 years
2. Type 2 diabetes mellitus (T2DM) or pre-diabetes, controlled by diet alone or metformin therapy and elevated blood pressure

   1. Pre-diabetes is defined as fasting plasma glucose of 100-125 mg/dL, plasma glucose of 140-199 mg/dL two hours after 75g oral glucose load, or hemoglobin A1C 5.7-6.4%. T2DM is defined as fasting plasma glucose of ≥126 mg/dL, plasma glucose of ≥200 mg/dL two hours after 75g oral glucose load, or hemoglobin A1C ≥6.5%.
   2. Elevated blood pressure is defined as systolic blood pressure (BP) ≥130 mmHg or diastolic BP ≥80 mmHg on three occasions or therapy with antihypertensive medication(s) for a minimum of three months.
3. For female subjects, the following conditions must be met:

   1. Postmenopausal status for at least one year or
   2. Status post-surgical sterilization, or
   3. If childbearing potential, utilization of birth control (barrier methods, abstinence, hormonal contraception, etc) and willingness to undergo regular beta hCG monitoring prior to drug treatment and on each study day. (Valsartan is pregnancy category D.)

Exclusion Criteria:

1. Type 1 diabetes
2. Poorly controlled T2DM, defined as hemoglobin A1C ≥8.7%
3. Use of anti-diabetic medications other than metformin for over 24 months prior to initiation of the study.
4. Requiring the need for insulin therapy
5. Secondary hypertension
6. Severe hypertension requiring the use of more than two anti-hypertensive agents other than a stable dose of diuretic or blood pressure > 180/110 mmHg
7. Subjects who have participated in a weight-reduction program during the last 6 months and whose weight has increased or decreased more than 5 kg over the preceding 6 months
8. Pregnancy or breastfeeding
9. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, angiotensin converting enzyme inhibitors, ARBs, or NEP inhibitors, as well as known or suspected contraindications to the study drugs
10. History of angioedema
11. History of pancreatitis or known pancreatic lesions
12. Clinically significant gastrointestinal impairment that could interfere with drug absorption
13. Significant cardiovascular disease such as myocardial infarction or cardiovascular surgery or angioplasty within six months prior to enrollment, presence of angina pectoris, arrhythmia with history of or risk of syncopal episodes or need for antiarrhythmic therapy, congestive heart failure (LV hypertrophy and diastolic dysfunction acceptable), deep vein thrombosis, pulmonary embolism, second- or third-degree AV block, mitral valve stenosis, hypertrophic cardiomyopathy, or coronary or carotid artery disease likely to require surgical or percutaneous intervention within six months of screening
14. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >3 x upper limit of normal range)
15. Impaired renal function (eGFR< 50mL/min/1.73m2 as determined by the MDRD equation)
16. History or presence of immunological or hematological disorders
17. Serum potassium >5.2 mmol/L at screening
18. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack within six months
19. Hematocrit <35%
20. Diagnosis of asthma requiring use of inhaled beta agonist more than once a week
21. Clinically significant gastrointestinal impairment that could interfere with drug absorption
22. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with daily use of non-steroidal anti-inflammatory drugs
23. Treatment with chronic systemic glucocorticoid therapy within the last year
24. Treatment with systemic glucocorticoid therapy acutely within six weeks prior to enrollment
25. Treatment with lithium salts
26. History of alcohol or drug abuse
27. Treatment with anticoagulation
28. Treatment with any investigational drug in the one month preceding the study
29. Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
30. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intact glucagon like peptide-1 (GLP-1) levels after the mixed meal | This will be measured just before the meal and after the meal at pre-specified time points for a total of four hours. (Time points 0 to 4 hours)
  GLP-1 is a hormone released after a meal that has been shown to improve insulin and glucose dynamics. It is a target for diabetes therapies. We will compare GLP-1 levels during the different drug treatments and at baseline.

SECONDARY OUTCOMES:
Insulin levels after the mixed meal | This will be measured just before the meal and after the meal at pre-specified time points for a total of four hours. (Time points 0 to 4 hours)
  Insulin is a hormone released from the pancreas that helps with blood glucose control. We will measure insulin levels during the different drug treatments and at baseline.
Blood glucose levels after the mixed meal | This will be measured just before the meal and after the meal at pre-specified time points for a total of four hours. (Time points 0 to 4 hours)
  We will compare blood glucose levels during the different drug treatments and at baseline.
Triglyceride levels after the mixed meal | This will be measured just before the meal and after the meal at pre-specified time points for a total of four hours. (Time points 0 to 4 hours)
  Triglycerides are a component of a routine lipid/ cholesterol panel. They rise in the setting of increased fat intake. GLP-1 is thought to decrease triglyceride levels. We will compare triglyceride levels during the different drug treatments and at baseline.
Neprilysin enzyme (drug) activity at baseline, during sacubitril/valsartan, and during valsartan | Time points -120 min (before drug given) and 0 min (2 hours after drug dose, just prior to the meal)
  Neprilysin is an enzyme that breaks down several proteins, including glucagon-like peptide-1 (GLP-1). Sacubitril in sacubitril/valsartan is a pro-drug of a neprilysin inhibitor. This assay level will help to determine if the changes seen after the meal are related to alterations in this enzyme activity and administration of the drug sacubitril/valsartan compared to valsartan. We will measure this before the medication is administered (thus at baseline) and two hours after the drug is administered and just prior to the mixed meal.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Wilson, MD, MSCI, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This study will not have large scale genomic data to share. The maximum number of participants will be 50.